CLINICAL TRIAL: NCT06222697
Title: Post Marketing Surveillance Study for Jivi (Damoctocog Alfa Pegol) in Korean Patients With Hemophilia A
Brief Title: A Study to Learn More About the Safety of Damoctocog-alfa-pegol When Used in Routine Medical Care in Korean Participants With Hemophilia A
Status: Recruiting | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 21278
Record Dates: First submitted 2023-12-19; First posted 2024-01-25 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Hemophilia A; Prophylaxis of Bleeding; Treatment of Bleeding
MeSH Terms: conditions — Hemophilia A | interventions — Factor VIII

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Post-marketing surveillance cohort: Participants follow their usual medical visits with data collection occurs continuously in a 36-week observational period.
  Interventions: Drug: Damoctocog-alfa-pegol (Jivi, BAY94-9027)

INTERVENTIONS:
Drug: Damoctocog-alfa-pegol (Jivi, BAY94-9027) — Follow clinical practice/administration. No drug is provided to participants due to the observational nature of the study.

SUMMARY:
In this study, researchers will observe and study the data from participants with hemophilia A who receive damoctocog alfa pegol as prescribed by their doctors. Participants will not receive any advice or changes to their healthcare during the study.

Hemophilia A is a genetic bleeding disorder. It is caused by the lack of a protein called clotting factor 8 (FVIII) that helps blood to clot properly. Lack of FVIII can result in excessive blood loss or bleeding inside the body after being injured or having surgery.

The study drug, damoctocog alfa pegol, can be used to prevent or treat bleeding episodes by replacing missing FVIII in the body of people with hemophilia A. It is already approved for people with hemophilia A who are at least 12 years old and have previously used other hemophilia A treatments.

Through this study, researchers want to learn more about its safety in a real-world setting.

The participants will receive damoctocog alfa pegol as prescribed by their doctors during routine practice according to the approved product information.

The main purpose of this study is to learn more about how safe damoctocog alfa pegol is in Korean participants with hemophilia A who previously used other hemophilia A treatments. To do this, researchers will collect information about any medical problems participants have during their treatment.

Data will be collected from December 2023 to March 2026 and cover a period of about 8 months for each participant. Data will come from participants' health records and information collected during their routine clinic visits.

In this study, only available data from routine care will be collected. No visits or tests are required as part of this study.

ELIGIBILITY:
Inclusion Criteria:

* ≥12 years of age with hemophilia A
* Previously treated with FVIII concentrate(s) (plasma derived or recombinant)
* Patients who have been treated with Jivi (damoctocog alfa pegol) and those for whom the decision to initiate treatment with Jivi was made as per physician's routine treatment practice with any kind of treatment modality (on-demand, prophylaxis, etc.)
* Written informed consent from subject or legal representative; assent from subject when appropriate

Exclusion Criteria:

* Contraindication according to the local authorized indication (including known hypersensitivity to the drug substance or any of its components (e.g., mouse or hamster protein))
* Patients participating in an investigational program with interventions outside of routine clinical practice
* Patients with any other diagnosis of bleeding/coagulation disorder other than hemophilia A
* Patients on immune tolerance induction treatment at the time of enrollment

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study should be conduct on hemophilia A patients who are prescribed with Jivi (damoctocog alfa pegol) as sole treatment for an approved indication (the treatment and prophylaxis of bleeding in PTPs aged ≥ 12 years with hemophilia A (congenital FVIII deficiency)) by the Ministry of Food and Drug Safety (MFDS) in Korea.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-01-24 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Occurrence of adverse events (AEs) | Up to 36 weeks
  Number of participants with AEs
Occurrence of Serious adverse events (SAEs) | Up to 36 weeks
  Number of participants with SAEs
Occurrence of adverse reactions (ARs) | Up to 36 weeks
  Number of participants with ARs
Occurrence of Serious adverse reactions (SARs) | Up to 36 weeks
  Number of participants with SARs
Occurrence of adverse events of important identified risks (AESIs) | Up to 36 weeks
  Important identified risks include development of Factor VIII inhibitors/Hypersensitivity/Clinical response characterised by lack of drug effect associated with anti-polyehtylene glycol (PEG) antibodies.
Number of adverse events related to overdose | Up to 36 weeks
Number of adverse events related to previously taken drugs and concomitant drugs | Up to 36 weeks

SECONDARY OUTCOMES:
Annualized number of reported total bleeds | Up to 36 weeks
Difference in annualized total number of injections, injection frequency from previous FVIII products versus Jivi (damoctocog alfa pegol) | Up to 36 weeks
Difference annualized total/average factor consumption (for overall, prophylaxis, bleeds(Intermittent prophylaxis), and other events) from previous FVIII products versus Jivi (damoctocog alfa pegol) | Up to 36 months
Regimen selection determinants (physician and patient) | Up to 36 weeks
Number of patients with 0 bleeds, and the difference in proportion comparing to previous prophylaxis treatment | Up to 36 weeks
ABR during the study compared with ABR for previous FVIII products in the 12 months prior to enrollment into the study | Up to 36 weeks
  ABR stands for annualized bleeding rate.

CONTACTS AND LOCATIONS:
Locations (1):
- Many Locations, Multiple Locations, South Korea

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.